CLINICAL TRIAL: NCT04227444
Title: Preoperative Evaluation of Pulmonary Vascular Anatomy by Augmented Reality (Holograms) in Patients Undergoing Lung Resection
Brief Title: Preoperative Evaluation of Pulmonary Vascular Anatomy by Holograms
Acronym: Holo-lungs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: R1033/19-IEO1088
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Disease; Lung Cancer
MeSH Terms: conditions — Lung Diseases; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hologram — Patient undergoing elective anatomical resection for lung cancer will receive standard preoperative CT scan of the chest (as usual); CT images will be subsequently elaborated by a Holographic computer to generate 3D images (holograms).Two radiologists and two thoracic surgeons will analyze CT images in a standard modality and report number of artery and vein branches for the lobe to be resected, moreover they will report every anatomical variation, according to the normal anatomy.
  After that, the same two radiologists and thoracic surgeons will analyze 3D images by the use of Microsoft Hololens and perform the same analysis as quoted above.
  For each review of the exam performed will be written a digitally signed clinical report to certify the timing of the evaluation and to be able to trace the analysis and any subsequent modifications of the interpretation of the CT images results.

SUMMARY:
Pulmonary vascular anatomy represents a constant challenge during lung resection, because of its variability in terms of vascular branches and anatomical variations.

Preoperative standard computed tomography is not always sufficient to foresee tricky abnormalities; augmented reality, thanks to holograms creation, may offer additional data on pulmonary vascular anatomy and its relation with neoplastic tissue. The aim of this study is to assess the possibility of correctly predict number, location and potential anomalies of pulmonary vascular anatomy of the lobe to be resected in patients undergoing lung resection for cancer.

Patients will receive standard preoperative oncologic and functional assessment. Preoperative computed tomography (CT) - performed according to a specific protocol - will be performed. CT images will be subsequently elaborated to generate 3D images (holograms). Two radiologists and two thoracic surgeons will analyze CT images and report number of artery and vein branches for the lobe to be resected. Moreover they will report every anatomical variation, according to the normal anatomy. After that, the same two radiologists and thoracic surgeons will analyze the holograms and perform the same analysis as quoted above. Patients will undergo to the planned surgical resection. The operating team will report the exact number of artery and vein branches of the resected lobe as well as every anatomical variation. Preoperative CT and holographic findings of the radiologists and the thoracic surgeons will be matched with the report of the operating team.

DETAILED DESCRIPTION:
An augmented reality (AR) system provides the surgeon with computer processed imaging data in real-time via dedicated hardware and software. The projection of AR is made possible by using displays, projectors, cameras, trackers, or other specialized equipment.

At present, the applications of AR are limited by the essential requisite of preoperative 3D reconstructions of medical images. It is possible to create these reconstructions by using commercial or self-made software from the Digital Imaging and Communications in Medicine (DICOM) format . The quality of a reconstruction depends on the quality of input data and the accuracy of the reconstruction system. Such reconstructions can be used for virtual exploration of target areas, planning an elective surgical approach in advance, and for better orientation and navigation in the operative ﬁeld. AR is especially useful in visualizing critical structures such as major vessels, nerves, or other vital tissues. By projecting these structures directly onto the patient, AR increases safety and reduces the time required to complete the procedure. Moreover Augmented reality proved to be an eﬀective tool for training and skill assessment of surgery residents, other medical staﬀ, or students. Augmented reality can be used eﬀectively for preoperative planning and completion of the actual surgery in timely fashion. The preoperative 3D reconstructed images can be modiﬁed and prepared for display in AR systems. Commonly, AR is used for tailoring individually preferred incisions and cutting planes, optimal placement of trocars, or to generally improve safety by displaying positions of major organ components. Another beneﬁt of AR is the ability to aid surgeons in diﬃcult terrain after a neoadjuvant chemotherapy or radiotherapy.

Studies suggest that AR systems are becoming comparable to traditional navigation techniques, with precision and safety suﬃcient for routine clinical practice. Most problems faced presently will be solved by further medical and technological research. Augmented reality appears to be a powerful tool possibly capable of changing the ﬁeld of surgery through a rational use. In the future, AR will likely serve as an advanced human-computer interface, working in symbiosis with surgeons, allowing them to achieve even better results. Nevertheless, further advancement is much needed to achieve maximum potential and cost-eﬀectiveness of augmented reality.

ELIGIBILITY:
Inclusion Criteria:

* Planned anatomical resection for lung cancer
* Signed and dated informed consent indicating that the patient has been informed of all pertinent aspects of the study.
* Willingness and ability to comply with study procedures.

Exclusion Criteria:

* Age younger than 18 years
* Contraindications to general anesthesia
* Poor general clinical conditions ( ECOG PS >=2)
* Patients unable to provide informed consent

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffering from (any) lung cancer scheduled for anatomical lung resection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Prediction of the exact number of pulmonary arteries and veins of the lobe to be resected. | 2020 - 2022
  Two different investigator (1 senior radiologist and 1 senior thoracic surgery) evaluate standard preoperative CT scan and indicate the number of pulmonary artery and veins of the lobe to be resected; this will be reported in a dedicated registry. After that, the same investigators will evaluate holograms of the same patients and will report the number of arteries and veins of the lobe to be resected; they will then register these data in the same registry. After the operation, the operating surgeon will report - as usual - the number of the arteries and veins resected during the procedure. Finally the prediction of the investigators obtained only by CT scan evaluation or bay CT scan + holograms evaluation, will be compared with the operatory report.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - European Institute of Oncology, Milan
  - European Institue of Oncology, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vavra P, Roman J, Zonca P, Ihnat P, Nemec M, Kumar J, Habib N, El-Gendi A. Recent Development of Augmented Reality in Surgery: A Review. J Healthc Eng. 2017;2017:4574172. doi: 10.1155/2017/4574172. Epub 2017 Aug 21. PMID 29065604
- [Background] Pessaux P, Diana M, Soler L, Piardi T, Mutter D, Marescaux J. Towards cybernetic surgery: robotic and augmented reality-assisted liver segmentectomy. Langenbecks Arch Surg. 2015 Apr;400(3):381-5. doi: 10.1007/s00423-014-1256-9. Epub 2014 Nov 13. PMID 25392120
- [Background] Inoue D, Cho B, Mori M, Kikkawa Y, Amano T, Nakamizo A, Yoshimoto K, Mizoguchi M, Tomikawa M, Hong J, Hashizume M, Sasaki T. Preliminary study on the clinical application of augmented reality neuronavigation. J Neurol Surg A Cent Eur Neurosurg. 2013 Mar;74(2):71-6. doi: 10.1055/s-0032-1333415. Epub 2013 Feb 12. PMID 23404553
- [Background] Pessaux P, Diana M, Soler L, Piardi T, Mutter D, Marescaux J. Robotic duodenopancreatectomy assisted with augmented reality and real-time fluorescence guidance. Surg Endosc. 2014 Aug;28(8):2493-8. doi: 10.1007/s00464-014-3465-2. Epub 2014 Mar 8. PMID 24609700
- [Background] Shakur SF, Luciano CJ, Kania P, Roitberg BZ, Banerjee PP, Slavin KV, Sorenson J, Charbel FT, Alaraj A. Usefulness of a Virtual Reality Percutaneous Trigeminal Rhizotomy Simulator in Neurosurgical Training. Neurosurgery. 2015 Sep;11 Suppl 3:420-5; discussion 425. doi: 10.1227/NEU.0000000000000853. PMID 26103444
- [Background] Lahanas V, Loukas C, Smailis N, Georgiou E. A novel augmented reality simulator for skills assessment in minimal invasive surgery. Surg Endosc. 2015 Aug;29(8):2224-34. doi: 10.1007/s00464-014-3930-y. Epub 2014 Oct 11. PMID 25303925
- [Background] Qu M, Hou Y, Xu Y, Shen C, Zhu M, Xie L, Wang H, Zhang Y, Chai G. Precise positioning of an intraoral distractor using augmented reality in patients with hemifacial microsomia. J Craniomaxillofac Surg. 2015 Jan;43(1):106-12. doi: 10.1016/j.jcms.2014.10.019. Epub 2014 Oct 29. PMID 25465484
- [Background] Muller M, Rassweiler MC, Klein J, Seitel A, Gondan M, Baumhauer M, Teber D, Rassweiler JJ, Meinzer HP, Maier-Hein L. Mobile augmented reality for computer-assisted percutaneous nephrolithotomy. Int J Comput Assist Radiol Surg. 2013 Jul;8(4):663-75. doi: 10.1007/s11548-013-0828-4. Epub 2013 Mar 23. PMID 23526436
- [Background] Volonte F, Pugin F, Bucher P, Sugimoto M, Ratib O, Morel P. Augmented reality and image overlay navigation with OsiriX in laparoscopic and robotic surgery: not only a matter of fashion. J Hepatobiliary Pancreat Sci. 2011 Jul;18(4):506-9. doi: 10.1007/s00534-011-0385-6. PMID 21487758
- [Background] Souzaki R, Ieiri S, Uemura M, Ohuchida K, Tomikawa M, Kinoshita Y, Koga Y, Suminoe A, Kohashi K, Oda Y, Hara T, Hashizume M, Taguchi T. An augmented reality navigation system for pediatric oncologic surgery based on preoperative CT and MRI images. J Pediatr Surg. 2013 Dec;48(12):2479-83. doi: 10.1016/j.jpedsurg.2013.08.025. PMID 24314190
- [Derived] Petrella F, Rizzo SMR, Rampinelli C, Casiraghi M, Bagnardi V, Frassoni S, Pozzi S, Pappalardo O, Pravettoni G, Spaggiari L. Assessment of pulmonary vascular anatomy: comparing augmented reality by holograms versus standard CT images/reconstructions using surgical findings as reference standard. Eur Radiol Exp. 2024 May 10;8(1):57. doi: 10.1186/s41747-024-00458-w. PMID 38724831